CLINICAL TRIAL: NCT03620812
Title: Influence of Rapeseed Proteins on the Postprandial Metabolic Response.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: UFOP Union for the promotion of oil and protein plants eV (Unknown); University of Halle Medical Faculty (Other)
Responsible Party: Principal Investigator, Ulf Schlegelmilch, Study Coordinator, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UFOP 062018
Record Dates: First submitted 2018-06-26; First posted 2018-08-08 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Health, Subjective
Keywords: rapeseed, protein, postprandial, glucose
MeSH Terms: interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rapeseed protein (Experimental): Three interventions are planned, in which the subjects will eat a test meal with added rape protein isolate (arm 1), a test meal with added soy protein isolate (arm 2) and a test meal without additional protein (arm 3) in random order on 3 days. The subjects are randomly assigned to one of the 3 treatment arms, ultimately resulting in 6 sequences (cross-over)
  Interventions: Dietary Supplement: rapeseed or soy protein or no protein
- soy protein (Active Comparator)
  Interventions: Dietary Supplement: rapeseed or soy protein or no protein
- no protein (Placebo Comparator)
  Interventions: Dietary Supplement: rapeseed or soy protein or no protein

INTERVENTIONS:
Dietary Supplement: rapeseed or soy protein or no protein — 25g rapeseed protein in comparison to 25g soy protein or no protein - dosage of 25 g per day

SUMMARY:
The aim of the study is to investigate the effect of rapeseed proteins on the postprandial metabolic response. Therefore, study participants will receive a meal rich in fat and carbohydrates with and without rapeseed protein or with soy protein that serves as control.

DETAILED DESCRIPTION:
The current study is a monocentric, controlled intervention study that will be conducted as cross-over design. Three interventions are planned and participants will be invited to consume a test meal with added rapeseed protein isolate, a test meal with added soy protein isolate and a test meal without additional protein. The evening before, the subjects will receive a standardized dinner. After a 12-hour fasting overnight, a cannula will be placed. Blood samples will be taken before and after eating the test meal rich in carbohydrate and fat. The test meal consists of pasta with oily tomato sauce with either 25 g of rapeseed protein, 25 g of soy protein or no additional protein. A total of 11 blood samples will be collected over a period of 6 hours. In the meantime, the blood pressure and pulse will be measured repeatedly and information on satiety will be recorded. The interventions will be interrupted by a period of, at least, 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women
* age between 18 and 65 years
* informed consent
* body mass index between 18,5 up to 29,9 kg/m2
* anamnesis without diagnostic findings

Exclusion Criteria:

* acute or chronic diseases ((hypertension, coronary diseases, renal diseases, diabetes, alcohol abuse etc.)
* intake of drugs (exemption: oral contraceptive)
* pregnancy or lactation
* food intolerance or allergies to mustard, soy, tomato, wheat
* participation on another trial
* blood donation - while last 2 month before the start of the study
* extensive physical activity (competitive sports, hard physical work)
* diet procedure
* smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-04-06 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
time course of glucose level | 0,15,30,45,60,90,120,180,240,300 and 360 min after ingestion of testmeal rich in carbohydrates and fat
  Impact of rapeseed protein on the postprandial blood glucose level

SECONDARY OUTCOMES:
Cholesterol | 0,15,30,45,60,90,120,180,240,300 and 360 min after ingestion of testmeal rich in carbohydrates and fat
  Impact of rapeseed protein on the postprandial levels of Cholesterol
triglycerides | 0,15,30,45,60,90,120,180,240,300 and 360 min after ingestion of testmeal rich in carbohydrates and fat
  Impact of rapeseed protein on the postprandial levels of triglycerides
short chain fatty acids | 0,15,30,45,60,90,120,180,240,300 and 360 min after ingestion of testmeal rich in carbohydrates and fat
  Impact of rapeseed protein on the postprandial levels of short chain fatty acids
indole-3-propionate | 0,15,30,45,60,90,120,180,240,300 and 360 min after ingestion of testmeal rich in carbohydrates and fat
  Impact of rapeseed protein on the postprandial levels of indole-3-propionate
amino acids | 0,15,30,45,60,90,120 and 180 min after ingestion of testmeal rich in carbohydrates and fat
  Impact of rapeseed protein on the postprandial levels of amino acids
hormones (insulin, ghrelin, FGF23) | 0,15,30,45,60,90,120,180,240,300 and 360 min after ingestion of testmeal rich in carbohydrates and fat
  Impact of rapeseed protein on the postprandial levels of hormones (insulin, ghrelin, FGF23)
time course of urea level, | 0,15,30,45,60,90,120,180,240,300 and 360 min after ingestion of testmeal rich in carbohydrates and fat
  Impact of rapeseed protein on the postprandial levels of urea
minerals and blood hsCRP | 0,15,30,45,60,90,120,180,240,300 and 360 min after ingestion of testmeal rich in carbohydrates and fat
  Impact of rapeseed protein on the postprandial levels of minerals and blood hsCRP
systolic and diastolic blood pressures | 0,15,30,45,60,90,120,180,240,300 and 360 min after ingestion of testmeal rich in carbohydrates and fat
  time course: measurement of blood pressure in mm Hg
feeling of satiety by means of a questionnaire | 0,15,30,45,60,90,120,180,240,300 and 360 min after ingestion of testmeal rich in carbohydrates and fat
heart rate | 0,15,30,45,60,90,120,180,240,300 and 360 min after ingestion of testmeal rich in carbohydrates and fat
  time course: measurement of heart rate in beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Stangl, Prof.Dr., Study Director — MLU, Institut für Agrar-und Ernährungswissenschaften
Locations (1):
- Martin-Luther-University Institute of Agriculture and Nutritional Science, Halle, Saxony-Anhalt, Germany